CLINICAL TRIAL: NCT04688580
Title: An Open-label, Crossover Study to Assess the Pharmacokinetics, Safety, and Tolerability of Various XW10172 Oral Immediate- and Modified-release Formulations in Healthy Adult Volunteers
Brief Title: Pharmacokinetics, Safety, and Tolerability of Various XW10172 Oral Formulations in Healthy Adult Volunteers
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: XWPharma (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: XW10172-102
Record Dates: First submitted 2020-11-14; First posted 2020-12-30 (Actual); Last update posted 2022-11-04 (Actual); Status verified 2022-11

CONDITIONS: Healthy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- XW10172 (Experimental)
  Interventions: Drug: XW10172

INTERVENTIONS:
Drug: XW10172 — Various formulations

SUMMARY:
The purpose of the study is to evaluate the safety, tolerability and pharmacokinetics of various formulations of XW10172 in healthy volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male of female participants who are 18 to 55 years of age, inclusive.
* Participant is willing and able to provide signed and dated written informed consent to participate prior to admission to the study.

Exclusion Criteria:

* Evidence or history of clinically significant gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, psychiatric, neurological, immunological, or endocrine disorders, poor vision, or allergic disease including drug allergies, including immediate type hypersensitivity. A history of childhood asthma that has resolved is acceptable.
* Participant who, for any reason, is deemed by the investigator to be inappropriate for this study; or has any condition which would confound or interfere with the evaluation of the safety, tolerability, pharmacokinetics or pharmacodynamics of the investigational drug; or is unable to comply with the study protocol.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 46 (Actual)
Dates: Start 2020-11-29 (Actual); Primary Completion 2021-12-14 (Actual); Study Completion 2021-12-14 (Actual)

PRIMARY OUTCOMES:
Maximum concentration (Cmax) | 12 hours
Trough concentration (Cmin) | 12 hours
Area under the concentration-time curve (AUC) from 0 to time of last quantifiable concentration (AUC0-tlast) | 12 hours
AUC from time 0 extrapolated to infinity (AUC0-inf) | 12 hours
AUC over the dosing interval (AUCtau) | 12 hours
Apparent terminal half-life (t1/2) | 12 hours
Cmax and AUC ratios of metabolite to XW10172 | 12 hours
Apparent oral clearance (CL/F) | 12 hours
Time to reach Cmax (Tmax) | 12 hours

SECONDARY OUTCOMES:
Incidence, severity, and causality of AEs | Up to 14 Days

CONTACTS AND LOCATIONS:
Overall Officials: Daniel M. Canafax, PharmD, Study Director — XWPharma
Locations (1):
- CMAX, Adelaide, South Australia, Australia